CLINICAL TRIAL: NCT06759974
Title: Prevalence of Accidental Awareness Under General Anesthesia in a University Hospital
Brief Title: Prevalence of AAGA
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assoc. Prof., Marmara University
Other Study IDs: 09.2024.1325
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Accidental Awareness During General Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Postoperative patients: The population will consist of patients receiving general anesthesia for elective surgery. Written informed consent will be obtained. A questionnaire will be administered to patients undergoing general anesthesia for elective surgery during the 2-24 hours in the postoperative period. Participants will report their experience with AAGA in the perioperative period through the Modified Brice questionnaire. The questionnaire is designed to determine the waking experiences under anesthesia and aims to comprehensively assess the feelings and thoughts that patients feel during this process. In addition, demographic information (age, gender, body mass index, etc.), clinical data (medical history, current health status, etc.), surgical and anesthesia-related information (type of surgery, anesthesia technique used, etc.) will be collected for each patient. These data will be used to identify differences between patients who develop AAGA and those who do not.

SUMMARY:
Accidental Awareness During General Anesthesia (AAGA) is a condition where patients regain partial or full consciousness during anesthesia, unable to move or react. This can lead to distressing experiences such as pain, fear, or stress, and may cause long-term psychological effects like insomnia, nightmares, and post-traumatic stress disorder. Although AAGA prevalence is reported as 0.1% to 0.2% in Western studies, data specific to populations like Turkey are limited and lack large-scale research. This study aims to investigate the prevalence of AAGA in Turkey and identify associated risk factors, including patient characteristics (e.g., age, gender, comorbidities), surgical variables, and anesthesia techniques. By addressing these factors, the study seeks to enhance anesthesia safety standards and provide critical data for national health policies and practices.

DETAILED DESCRIPTION:
Accidental Awareness During General Anesthesia (AAGA) is defined as a state in which the patient accidentally gains partial or full consciousness during anesthesia and is unable to move or react. This state is often associated with uncomfortable sensations in the patient, such as pain, fear and intense stress during the operation. Awareness is a serious condition that causes anxiety in patients, even if they do not feel any pain. These patients may experience insomnia, recurrent nightmares and post-traumatic stress disorder in the postoperative period. The prevalence and long-term effects of AAGA are of great importance for the safety of anesthesia practices.

In the available literature, the prevalence of AAGA in patients under general anesthesia has been reported as 0.1% to 0.2%. However, since these data are generally based on European and American populations, comprehensive studies in different populations such as Turkey are needed. Studies in Turkey usually have limited sample sizes. This study aims to better understand the prevalence of AAGA in Turkey and to provide important information to contribute to national health policies and anesthesia practice.

In this study, the prevalence of AAGA will be determined and its relationship with patient, surgical and anesthesia factors will be investigated. Determining the risk factors of AAGA is critical for patient safety and is expected to vary in different patient cohorts. In particular, variables such as age, gender, comorbidity, type and duration of anesthesia used are thought to be factors that play a role in the occurrence of AAGA. Moreover, it is suggested that different types and durations of surgery may also affect the risk of AAGA.

This study is expected to contribute to the improvement of safety standards under general anesthesia and to fill the data gap in the national literature by analyzing the prevalence and risk factors of AAGA in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia under elective conditions
* American Society of Anesthesiologists (ASA) physical status I-III patients

Exclusion Criteria:

* Patients who are not capable of understanding and analyzing the test
* Patients with neurodegenerative diseases such as dementia, Alzheimer's disease
* Patients not extubated in the postoperative period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study will consist of adult patients receiving general anesthesia for elective surgery at Marmara University Pendik Training and Research Hospital and Prof. Dr. Asaf Ataseven Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2546 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Accidental Awareness During General Anesthesia, AAGA | During the 2-24 hours postoperatively.
  Experience of the Accidental Awareness During General Anesthesia in the early perioperative period that will be obtained via a questionnaire during the postoperative day zero.

IPD SHARING:
Plan to Share IPD: Undecided